CLINICAL TRIAL: NCT02591199
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Multi-Center Single Dose Study to Evaluate the Safety and Effectiveness of URG101 Compared With the Individual Components Lidocaine and Heparin in Subjects With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Engage 24: Evaluation of the Safety and Effectiveness of URG101 in Subjects With Interstitial Cystitis/Bladder Pain Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely terminated due to data inconsistent with the experimental plan and lack of funding
Sponsor: Urigen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URG101-105
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Lidocaine; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- URG101 (Experimental): A single 15 mL dose of URG101,a mix of buffered Lidocaine (200 mg) and Heparin (50,000 IU), delivered to the bladder via catheter.
  Interventions: Drug: URG101
- Placebo (Placebo Comparator): A single 15 mL dose of placebo delivered to the bladder via catheter.
  Interventions: Drug: Placebo
- Lidocaine (Experimental): A single 15 mL dose of buffered Lidocaine (200 mg) delivered to the bladder via catheter.
  Interventions: Drug: Lidocaine
- Heparin (Experimental): A single 15 mL dose of buffered Heparin (50,000 IU) delivered to the bladder.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: URG101
  Arms: URG101
Drug: Placebo
  Arms: Placebo
Drug: Lidocaine
  Arms: Lidocaine
Drug: Heparin
  Arms: Heparin

SUMMARY:
The purpose of this study is to determine if the combination product (URG101) is safe and effective versus its individual components (Heparin Sodium and Lidocaine Hydrochloride) for the treatment of Interstitial Cystitis/Bladder Pain Syndrome. The study is randomized and double-blinded such that neither the subject nor doctor will know which drug or placebo is received.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo controlled, multicenter, single-dose, pharmacokinetic study designed to determine the efficacy and safety of the combination product (URG101) compared with its individual components (Heparin Sodium and Lidocaine Hydrochloride).

Eligible subjects exhibiting moderate to severe symptoms of bladder pain associated with their diagnosis of interstitial cystitis/bladder pain syndrome who have signed informed consent, will be screened and provisionally enrolled for intravesical treatment.

On the day of study drug administration subjects will be randomized (2:1:2:1; URG101:placebo:lidocaine:heparin) and will receive a single administration of one of four intravesical treatments in a blinded fashion, based on random assignment:

1. URG101 (buffered lidocaine-heparin)
2. Placebo (phosphate buffer)
3. Lidocaine hydrocholoride buffered alone
4. Heparin sodium buffered alone

Efficacy and safety assessments will be completed for 24 hours after study drug administration. End of Study Follow-up will be completed by telephone 48 to 72 hours after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

Subjects diagnosed with interstitial cystitis/bladder pain syndrome must meet all of the following criteria to participate in the study:

1. Have provided written informed consent to participate in this trial
2. Be male or female, ≥ 18 years of age
3. Have moderate-to-severe symptoms of bladder pain of bladder origin for at least 9 months prior to the study
4. May or may not have received a cystoscopy in association with their diagnosis of interstitial cystitis/bladder pain syndrome prior to or at time of screening
5. Have a score of ≥ 15 and < 30 on the PUF questionnaire, completed at screening
6. A minimum score of 5 is required on the VAS
7. Have been using a stable dose of hormone therapy for ≥ 3 months, if female and currently taking hormone therapy

Exclusion Criteria:

1. Pregnant or breastfeeding. For females of child bearing potential and males, if sexually active, must be willing to commit to an acceptable method of birth control for the duration of the study.
2. Have a known hypersensitivity to heparin or lidocaine
3. Have used any local anesthetic by any route within 24 hours prior to study drug administration, or used a lidocaine patch within 14 days prior to study drug administration
4. Have used a tricyclic antidepressant or a gamma-Aminobutyric acid (GABA) analogue (gabapentin or pregabalin) unless taking the medication for ≥ 3 weeks. The stable dose of gabapentin may not exceed 1,200 mg per day, and the stable dose of pregabalin may not exceed 150 mg per day.
5. Have used any pain medication within 6 hours prior to study drug administration
6. Have used narcotics or medical marijuana ≤ 3 weeks prior to study entry (generic names: fentanyl, hydrocodone, hydromorphone, levorphanol, medical marijuana, methadone, morphine, oxycodone, propoxyphene, tramadol). Subjects who have received codeine within this time period may be admitted if the use is not chronic, and not within 6 hours of enrollment, such that they are not at risk for GI or opiate withdrawal symptoms that in the opinion of the investigator would impact the subject's study participation due to their ability to follow the study protocol or bias study results.
7. Have used prohibited drugs as determined by self-report, positive urine drug screen, or in the opinion of the investigator be under the influence of drugs affecting mentation precluding their ability to follow the study protocol or bias study results
8. Have a known clinically significant abnormal laboratory test value defined by the investigator
9. Have a neurogenic bladder or other disorder that, in the opinion of the investigator, may cause neurogenic bladder (including Parkinson's disease, multiple sclerosis, epilepsy, myasthenia gravis, movement disorders, spinal cord damage)
10. Have pain or a pain disorder that, in the opinion of the investigator, would make it difficult to discriminate pelvic pain of bladder origin from the other pain
11. Have severe depression, bipolar disorder, schizophrenia, anxiety, attention deficit disorder, obsessive compulsive disorder, or other major central nervous system disorder
12. Have history of arrhythmias, conduction disturbances, or cardiac disease, or any coexisting medical condition that, in the opinion of the investigator, may be significant or interfere with study procedures or interpretation of study results
13. Had bladder instillation therapy within 7 days prior to study entry or had a prior bladder instillation with heparin and lidocaine and did not respond
14. Had dilatation (hydrodistention) of bladder within 3 months of study entry
15. Evidence or suspected presence of cancer detected during cystoscopy prior to or at time of initial screening.
16. Has received any investigational drug or device within 30 days prior to screening
17. Is currently enrolled in another investigational drug or device study
18. Is unwilling or unable to abide by the requirements of the study
19. Have an actively bleeding lesion or area in the bladder as detected by dipstick urinalysis and investigator assessment, immediately prior to randomization
20. Have had any of the following: bacterial, chemical (including ketamine and cyclophosphamide) or radiation cystitis; gynecological, urological or rectal cancer; current chemotherapy; tuberculous cystitis; urinary schistosomiasis; bladder or uretal calculi; vaginitis or genital herpes; urethral diverticulum or bladder fistulae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-09; Primary Completion 2018-05-14 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Lowell Parsons, MD, Study Chair — Urigen
Locations (11):
- United States (11):
  - IC Study, LLC, Escondido, California
  - University of California San Diego, San Diego, California
  - Georgia Urology, Cartersville, Georgia
  - The Urogynecology Center, Overland Park, Kansas
  - Rutgers Women's Health Clinic, New Brunswick, New Jersey
  - The Arthur Smith Institue for Urology- North Shore Long Island Jewish Health System, Lake Success, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - MetroHealth System, Center for Advanced Gynecology, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - Urology of Virginia, PLLC, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- URG101: A single 15 mL dose of URG101,a mix of buffered Lidocaine (200 mg) and Heparin (50,000 IU), delivered to the bladder via catheter.
  URG101
- Heparin: A single 15 mL dose of buffered Heparin (50,000 IU) delivered to the bladder.
  Heparin
- Lidocaine: A single 15 mL dose of buffered Lidocaine (200 mg) delivered to the bladder via catheter.
  Lidocaine
- Placebo: A single 15 mL dose of placebo delivered to the bladder via catheter.
  Placebo
Period: Overall Study
Arm/Group | URG101 | Heparin | Lidocaine | Placebo
Started | 31 | 15 | 29 | 16
Completed | 31 | 15 | 29 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | URG101 | Heparin | Lidocaine | Placebo | Total
Number analyzed (Participants) | 31 | 15 | 29 | 16 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (15.06) | 52.2 (16.86) | 45.3 (15.41) | 50.2 (16.15) | 47.8 (15.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 14 | 28 | 13 | 85
  Male | 1 | 1 | 1 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 5 | 4 | 15
  Not Hispanic or Latino | 26 | 14 | 24 | 12 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 0 | 1 | 8
  White | 27 | 8 | 28 | 15 | 78
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average of Bladder Sum of Pain Intensity Differences From Baseline to 12 Hours (SPID-12) as Determined Using an 11-point Numeric Rating Scale (NRS) for Pain Intensity
Description: A calculation of average bladder Sum of Pain Intensity Differences from Baseline to 12 hours (SPID-12). A pain intensity score of 0 (no pain) to 10 (worst possible pain) is obtained before starting the study and throughout the 12 hour time period. The average SPID-12 is calculated by multiplying the Pain Intensity Difference score at each time point by the duration since the preceding time point and then summing these values over the specific time period. A lower, negative average SPID-12 difference is better and indicates a reduction in pain intensity compared to the baseline score, whereas a positive score indicates an increase in pain intensity compared to baseline. The full range of results of the average SPID-12 difference could be -119 to +59.
Time Frame: 12 hours
Population: Subjects included in this analysis must have received a dose of the applicable study treatment and completed through the 12 hour SPID collection timepoint. Intent to Treat / Safety Population includes all subjects who received the relevant dose; Per Protocol Population includes all subjects who met entrance criteria; Per Protocol Instillation History includes a subset of the Per Protocol Population who previously received at least one instillation treatment.
Measure: Mean (Standard Deviation); unit: units on a scale*hours
Arm/Group | URG101 | Heparin | Lidocaine | Placebo
Number analyzed (Participants) | 31 | 15 | 29 | 16
units on a scale*hours
  Intent to Treat / Safety Population | -30.81 (21.641) | -22.50 (25.918) | -27.50 (26.121) | -19.63 (18.558)
  Per Protocol Population: number analyzed (Participants) | 28 | 14 | 27 | 13
  Per Protocol Population | -33.41 (20.89) | -24.11 (26.11) | -26.43 (26.76) | -15.42 (17.74)
  Per Protocol-Instillation (history of receiving bladder instillations) Population: number analyzed (Participants) | 19 | 8 | 14 | 10
  Per Protocol-Instillation (history of receiving bladder instillations) Population | -37.51 (18.06) | -12.38 (22.38) | -23.27 (25.96) | -16.28 (19.66)

2. Primary Outcome: Change of Bladder Sum of Pain Intensity Differences From Baseline to 12 Hours (SPID-12) as Determined Using an 11-point Numeric Rating Scale (NRS) for Pain Intensity
Description: A calculation of bladder Sum of Pain Intensity Differences from Baseline to 12 hours (SPID-12) after administration of URG101 compared with the SPID-12 after administration of lidocaine alone, heparin alone, and placebo. A pain intensity score of 0 (no pain) to 10 (worst possible pain) is obtained before starting the study and throughout the 12 hour time period. A negative value indicates lower SPID-12 values for URG101. The full range of results of the average SPID-12 difference could be -119 to +59.
Time Frame: 12 hours
Population: Overall numbers of participants reflects all participants who received at least one dose of study drug (URG101), comparators (Heparin or Lidocaine), or placebo. The above arm numbers compare URG101 to its individual components of heparin, lidocaine, and placebo, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale*hours
Groups:
- URG101 Minus Heparin: Comparison of least squares mean difference of bladder sum of pain intensity scores (SPID-12) for URG101 minus Heparin
- URG101 Minus Lidocaine: Comparison of least squares mean difference of bladder sum of pain intensity scores (SPID-12) for URG101 minus Lidocaine
- URG101 Minus Placebo: Comparison of least squares mean difference of bladder sum of pain intensity scores (SPID-12) for URG101 minus Placebo
Arm/Group | URG101 Minus Heparin | URG101 Minus Lidocaine | URG101 Minus Placebo
Number analyzed (Participants) | 46 | 60 | 47
units on a scale*hours
  Intent-to-Treat / Safety Population | -11.65 [-25.61 to 2.31] | -4.31 [-16.00 to 7.38] | -12.46 [-26.59 to 1.68]
  Per Protocol Population: number analyzed (Participants) | 42 | 55 | 41
  Per Protocol Population | -15.69 [-29.57 to -1.81] | -9.21 [-21.13 to 2.72] | -21.28 [-36.07 to -6.49]
  Per Protocol-Instillation (history of receiving bladder instillations) Population: number analyzed (Participants) | 27 | 33 | 29
  Per Protocol-Instillation (history of receiving bladder instillations) Population | -26.02 [-43.62 to -8.43] | -14.64 [-31.47 to 2.20] | -26.04 [-44.07 to -8.01]

ADVERSE EVENTS:
Time Frame: From the time of study drug administration through 72 hours post-dose
Arm/Group | URG101 | Heparin | Lidocaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/15 | 0/29 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/15 | 0/29 | 0/16
Other Adverse Events (participants affected / at risk) | 3/31 | 1/15 | 5/29 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | URG101 (N=31) | Heparin (N=15) | Lidocaine (N=29) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vertigo (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 2 | 1
Burning in Bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pain with Urination (Renal and urinary disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The IDMC reported a trend toward significance for URG101; but it was determined that >300 subjects would be required to reach significance. The data showed inconsistencies between different sites that could affect the ability to pool the data and could not be explained in a blinded analysis. Therefore, at 92 subjects enrolled, the study was terminated early due to data inconsistent with the experimental plan, lack of funding. There is no SAP. Results are limited to primary endpoint and safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT02591199/Prot_SAP_000.pdf